CLINICAL TRIAL: NCT00782314
Title: Evaluating the Symbicort Turbuhaler (Formoterol/Budesonide) Maintenance and Reliever Therapy for Asthma in Daily Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Meta Jeras, Mr Ph, Regulatory and Medical Affairs Manager, AstraZeneca UK Limited, Branch Office in Slovenia
Other Study IDs: NIS-RSI-SYM-2008/1
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: asthma; SMART; Symbicort Turbuhaler; asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with maintenance only treatment with Symbicort Turbuhaler for at least 1 month
- 2: patients with SMART treatment with Symbicort Turbuhaler for at least 1 month

SUMMARY:
We want to evaluate efficacy of Symbicort® Turbuhaler® (formoterol/budesonide) therapy for asthma in real life conditions. For this purpose we will include both patients that are treated with Symbicort® Turbuhaler® the "classical" maintenance only treatment approach as well as those treated with the SMART approach.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with persistent asthma treated with Symbicort® Turbuhaler® in line with its label
* non-pregnant females
* existing maintenance only treatment with Symbicort® Turbuhaler® 80 μg/4,5 μg, 160 μg/4,5 μg or 320 μg/9 μg for at least 1 month
* existing SMART treatment with Symbicort® Turbuhaler® 80 μg/4,5 μg or 160 μg /4,5 μg for at least 1 month

Exclusion Criteria:

* patients not being treated with Symbicort® Turbuhaler®
* patients treated with Symbicort® Turbuhaler® for COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients visiting pulmologist's office
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-04; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
to determine the efficacy of both possible treatment approaches with Symbicort® Turbuhaler®, measured by asthma control | three times: 0, 3, 6 months after inclusion

SECONDARY OUTCOMES:
to determine the number of maintenance and reliever inhalations of Symbicort® Turbuhaler®, as well as the concomitant usage of a separate reliever inhaler even in the case of SMART treatment approach | three times: 0, 3, 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Igor Koren, MD, MSc, Principal Investigator — Radix - medicinske storitve, Igor Koren s.p.
Locations (24):
- Slovenia (24):
  - Research Site, Celje, Celje
  - Research Site, Dvorec Sela, Dvorec Sela
  - Research Site, Grosuplje, Grosuplje
  - Research Site, Idrija, Idrija
  - Research Site, Izola, Izola
  - Research Site, Jesenice, Jesenice
  - Research Site, Kamnik-Duplica, Kamnik-Duplica
  - Research Site, Kranj, Kranj
  - Research Site, Litija, Litija
  - Research Site, Ljubljana, Ljubljana
  - Research Site, Lucija, Lucija
  - Research Site, Maribor, Maribor City Municipality
  - Research Site, Novo Mesto, Mestna Občina Novo mesto
  - Research Site, Murska Sobota, Murska Sobota
  - Research Site, Domžale, Občina Domžale
  - Research Site, Ravne na Koroškem, Občina Ravne na Koroškem
  - Research Site, Sežana, Občina Sežana
  - Research Site, Ptuja, Ptuja
  - Research Site, Slovenj Gradec, Slovenj Gradec
  - Research Site, Slovenska Bistrica, Slovenska Bistrica
  - Research Site, Topolšica, Topolsica
  - Research Site, Velenje, Velenje
  - Research Site, Vrhnika, Vrhnika
  - Research Site, Zagorje, Zagorje